CLINICAL TRIAL: NCT03444142
Title: Effect of the Weekly Administration of Exenatide LAR or Dulaglutide on the Variability of Blood Pressure and Heart Rate of 24 Hours in Patients With Type 2 Diabetes Mellitus Without Pharmacological Treatment.
Brief Title: Effect of Exenatide LAR or Dulaglutide on the Variability of 24-hour Heart Rate and Blood Pressure in Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exenatida LAR Dulaglutida-with
Record Dates: First submitted 2018-02-13; First posted 2018-02-23 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Hyperglycemia; ABPM; Variability of blood pressure; Exenatide LAR or Dulaglutide 0.75mg; Glucagon-like peptide analogues type 1 (GLP1).
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia | interventions — Exenatide; dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Exenatide LAR (Active Comparator): Exenatide LAR 2 mg, once weekly subcutaneously before breakfast during 4 weeks.
  Interventions: Drug: Exenatide LAR
- Drug: Dulaglutide (Active Comparator): Dulaglutide .75 mg, once weekly subcutaneously Before breakfast during 4 weeks.
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Exenatide LAR — 2 mg, once weekly subcutaneously before breakfast during 4 weeks.
  Other Names: Bydureon
  Arms: Drug: Exenatide LAR
Drug: Dulaglutide — .75 mg once weekly subcutaneously before breakfast during 4 weeks.
  Other Names: Trulicity
  Arms: Drug: Dulaglutide

SUMMARY:
Mortality due to cardiovascular problems is increased by having Diabetes Mellitus type 2 (DM2), related to the time of evolution and glucose levels or if alterations in blood pressure coexist. With this variability there is greater damage to the target organ and in patients with DM2 the process is more severe and frequent due to alterations in the coagulation mechanisms that accelerate in the presence of hypertension, figures ≥135 / 85 mmHg are considered risk factors to develop coronary, cerebral or renal events. As a quantitative range, blood pressure is currently monitored ambulatory by (MAP) which is the most used and reliable non-invasive instrument for its evaluation. The American Association of Clinical Endocrinologists (AACE) proposes an algorithm that contemplates initiating management to patients with a diagnosis of diabetes with drugs such as metformin, thiazolidinediones and glucagon-like peptide analogues type 1 (GLP1).

Exenatide LAR and Dulaglutide are GLP-1 analogue drugs with potential to decrease the progressive losses of pancreatic β cell function and mass and cardiovascular risk (CV) factors with maintained use, in addition to hypoglycemic, hypotensive effects, weight decreases and visceral adiposity, however, it has been reported that although they share the same basic mechanism of action, each one has a different molecular structure and pharmacokinetic profile that make their pharmacological and clinical effects different, in particular as regards the variability of blood pressure and heart rate.

DETAILED DESCRIPTION:
A randomized, open clinical trial of 30 patients with a diagnosis of diabetes in accordance with the American Diabetes Association (ADA) without treatment.

They will be assigned randomly in two groups of 15 patients each to receive 2 mg subcutaneous of Exenatide LAR (Bydureon by Astra Zeneca) or Dulaglutide .75 mg (trulicity, by Lilly), once weekly before breakfast during 4 weeks.

There will be calculated body mass index (BMI); low-density lipoprotein cholesterol (LDL-c); very-low density lipoprotein (VLDL), glomerular filtration rate and blood pressure variability. This protocol it's already approved by the local ethics committee with number CEI/447/2017 and written informed consent it's going to be obtained from all volunteers.

Statistical analysis will be presented through measures of central tendency, dispersion, average and deviation standard for quantitative variables, frequencies and percentages for variable qualitative. Qualitative variables will be analyzed by X2, will be used for differences inter-group Mann-Whitney U Test and Wilcoxon Test for the within-groups differences. It will be considered statistical significance p ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 31 and 60 years
* Diagnosis of diabetes according ADA criteria:

(Fasting blood glucose levels >125 mg/dl or postprandial blood glucose levels after an oral glucose tolerance test with 75 of oral glucose > 200 mg/dl, or glycosylated hemoglobin >6.5%).

• Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to ingredients of intervention
* Physical impossibility for apply the drug
* Known pancreatic, renal, hepatic, heart or thyroid diseased
* Hypertension diagnosis
* Previous treatment for glucose
* Body Mass Index ≥39.9 kg/m2
* Triglycerides ≥500 mg/dL
* Total cholesterol ≥300 mg/dL
* Night or rotating shift workers
* Blood Pressure ≥140/90 mmHg

Ages: 31 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-17 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate: nighttime, daytime and 24-h | Baseline to Week 4
  heart rate variability will be evaluated with ambulatory blood pressure monitoring (ABPM) for 24 h by oscillometric method Microlife WatchBP O3
Systolic blood pressure, daytime, night and 24 h | Baseline to Week 4
  Blood pressure variability will be evaluated with ambulatory blood pressure monitoring (ABPM) for 24 h by oscillometric method Microlife WatchBP O33.
Diastolic blood pressure, daytime, night and 24 h | Baseline to Week 4
  Blood pressure variability will be evaluated with ambulatory blood pressure monitoring (ABPM) for 24 h by oscillometric method Microlife WatchBP O3
Blood pressure | Baseline to Week 4
  Blood pressure will be measured at baseline and week 4 with a digital sphygmomanometer and the entered values reflect the blood pressure.

SECONDARY OUTCOMES:
Categories: dipper o non dipper | Baseline to Week 4
  Blood pressure variability will be evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hrs by oscillometric method Microlife WatchBP O3
Fasting glucose levels | Baseline to Week 4
  The fasting glucose levels will be evaluated at baseline and week 4 with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at week 4
Central and peripheral blood pressure | Baseline to Week 4
  To determine and compare the effect of administration of Exenatide LAR or Dulaglutide on Central and peripheral blood pressure through HEM will be evaluated at baseline and week 4.
Pulse wave velocity | Baseline to Week 4
  To determine and compare the effect of administration of Exenatide LAR or Dulaglutide on pulse wave velocity through VP1000-plus with Ankle-Brachial Index will be evaluated at baseline and week 4.
Cardio-ankle Vascular Index (CAVI) | Baseline to Week 4
  To determine and compare the effect of administration of Exenatide LAR or Dulaglutide on arterial stiffness through Cardio-ankle Vascular Index (CAVI) will be evaluated at baseline and week 4.
Glycosylated hemoglobin | Baseline to Week 4
  Glycosylated hemoglobin will be evaluated at baseline and week 4 by high pressure liquid chromatography (HPLC) and the entered values reflect the glycosylated hemoglobin at week 4
Body Weight | Baseline to Week 4
  The body weight will be measured at baseline and week 4 with a bioimpedance balance and the entered values reflect the body weight at week 4
Body Mass Index | Baseline to Week 4
  Body Mass Index will be calculated at baseline and week 4 with the Quetelet index formula and the entered values reflect the body mass index at week 4
Total cholesterol | Baseline to Week 4
  Total cholesterol levels will be evaluated at baseline and week 4 by enzymatic/colorimetric techniques and the entered values reflect the total cholesterol level at week 4
Triglycerides levels | Baseline to Week 4
  Triglycerides levels will be evaluated at baseline and week 4 with enzymatic/colorimetric techniques and the entered values reflect the triglycerides level at week 4
High density lipoprotein (c-HDL) levels | Baseline to Week 4
  c-HDL levels will be evaluated at baseline and week 4 with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at week 4
Alanine aminotransferase (ALT) levels | Baseline to Week 4
  ALT levels will be evaluated at baseline and week 4 with enzymatic/colorimetric techniques
Aspartate aminotransferase (AST) levels | Baseline to Week 4
  AST levels will be evaluated at baseline and week 4 with enzymatic/colorimetric techniques [Time Frame: Baseline to Week 4
Creatinine levels | Baseline to Week 4
  Creatinine levels will be evaluated at baseline and week 4 with enzymatic/colorimetric techniques
Uric acid levels | Baseline to Week 4
  Uric acid levels will be evaluated at baseline and week 4 with enzymatic/colorimetric techniques
Waist Circumference | Baseline, week 4
  Waist circumference will be evaluated at baseline and at week 4 with a flexible tape

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de terapeutica Experimental y Clinica. Centro universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico